CLINICAL TRIAL: NCT05426954
Title: Blood Flow Restrictive Training Following Medial Patellofemoral Ligament and Anterior Cruciate Ligament Reconstruction Rehabilitation
Brief Title: BFRT MPFL and ACL Reconstruction Rehab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Richard Watson, PT (Other)
Responsible Party: Sponsor-Investigator, Richard Watson, PT, Co-Invetigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 54653
Record Dates: First submitted 2022-06-02; First posted 2022-06-22 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Medial Patellar Femoral Ligament Reconstruction Rehabilitation; Anterior Cruciate Ligament Reconstruction Rehabilitation
Keywords: rehabilitation

STUDY DESIGN:
Intervention Model Description: Randomized Rehabilitation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BFR deflate (Active Comparator): BFR cuff will be deflated at the end of each of the 4 BFR exercises, BFR cuff is inflated prior to start next BFR exercise.
  Interventions: Other: Rehabilitation utilizing blood flow restrictive therapy
- BFR do not deflate (Active Comparator): BFR cuff will not be deflated at the end of each of the 4 BFR exercises. Cuff remains inflated start exercise 1 thru completion exercise 4.
  Interventions: Other: Rehabilitation utilizing blood flow restrictive therapy

INTERVENTIONS:
Other: Rehabilitation utilizing blood flow restrictive therapy — BFR therapy

SUMMARY:
Blood flow restrictive (BFR) therapy following MPFL or ACL reconstruction rehabilitation.

Specific Aim 1: Test whether maintaining BFR cuff inflation or deflating between exercises results in greater quadriceps strength and functional outcomes after MPFL or ACL reconstruction.

Hypothesis 1: Subjects in the deflate BFR protocol group will have significantly greater quadriceps strength, symmetric leg symmetry index on a battery of functional tests and PROs as compared to the non-deflate group.

Specific Aim 2: Compare whether maintaining BFR cuff inflation or deflating between exercises results in reduced pain, improved exercise tolerance, and patient-reports outcomes (PRO) after MPFL or ACL reconstruction.

Hypothesis 2: Subjects in the deflated BFR protocol group will report significantly less pain and greater exercise tolerance during exercise with significantly improved knee related PRO scores.

DETAILED DESCRIPTION:
Subjects will be aged 13-40 male or female patient following MPFL or ACL reconstruction.

Baseline Assessment at PT Evaluation will included knee AROM and AAROM Heel slide with strap, Knee edema measured in cm difference Involved to Non-involved at supra and mid patellar levels, subjects ability to SLR Yes/No in brace, Patient reported outcome measure (PRO's) to include LEFS, Brief Resiliency scale, MPFL - Norwich Patellar instability, ACL 2000 IKDC Subjective Knee Evaluation Form questionnaires. Pain assessment to include current, minimal and maximal pain levels past 24 hours.

Patient are randomized into 1 of 2 groups: Group 1 will deflate between BFR exercises, Group 2 will not deflate between BFR exercises. Both groups will receive the same standard care same during their first 2 weeks of post-op rehabilitation. BFR will be added to their rehabilitation care starting at week 3 for 2x/week x 10. There are 4 core BFR exercises that will be progressed every 2 weeks.

Final Assessment- Strength and Functional Testing at 24th visit or 12 weeks post-op (if missed appointments) to include bilateral Knee AROM and edema assessments, PRO's: LEFS, Brief Resiliency scale, MPFL Norwich Patellar instability, ACL 2000 IKDC Subjective Knee Evaluation Form, Functional assessment to include for involved adn uninvolved leg: Isometric Quad strength measurement at 90 degrees of knee flexion, Isometric Hip Abduction strength measurement, Y balance maximum anterior reach, Max reps 6" Forward step-down, max core strength assessments, and ability in-line jog.

ELIGIBILITY:
Inclusion Criteria:

Post operative Medial Patellar Femoral Ligament or Anterior Cruciate Ligament Reconstruction.

Exclusion Criteria:

* Had any other previous surgeries or conditions that might affect your gait prior to injury and 1 year removed from a prior ACL or MPFL reconstruction.
* Have any current lower extremity condition other than MPFL or ACL reconstruction which might affect your gait
* Have a diminished capacity to provide informed consent
* Are diabetic or have uncontrolled hypertension
* Have recent inflammation, bleeding disorders, active bleeding or infection within the lower limbs.
* You are taking warfarin/Coumadin, clopidogrel/Plavix, Rivaroxaban/Xarelto, Dabigatran/Pradaxa, apixaban/Eliquis, deoxidant/Savaysa, betrixaban, or any other anti-coagulants that may cause excess bleeding.
* Have any implanted medical device
* Have a history of deep vein thrombosis, vascular graft, varicose veins, and/or sickle cell anemia
* Are or suspect you are Pregnant
* You are not be able to attend regular physical therapy or study visits

Ages: 13 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
Quadriceps Isometric Knee Strength | 24th visit or 12 weeks Post-op (if missed appointments)
  involved vs uninvolved isometric quadriceps knee strength measured at 90 degrees flexion comparison
Hip abduction Isometric Strength | measured at the 24th visit or 12 weeks Post-op (if missed appointments)
  involved vs uninvolved isometric hip abduction strength comparison
Y Balance Anterior Reach Test | measured at the 24th visit or 12 weeks Post-op (if missed appointments)
  involved vs uninvolved maximum Y Anterior Reach test comparison
Maximum 6 inch forward step down test | measured at the 24th visit or 12 weeks Post-op (if missed appointments)
  involved vs uninvolved maximum reps performing 6" forward step down in 1 min comparison
Max core strength assessment | measured at the 24th visit or 12 weeks Post-op (if missed appointments)
  Max hold in seconds: prone plank, side planks and single leg bridge
Ability to in-line jog | measured at the 24th visit or 12 weeks Post-op (if missed appointments)
  Determine if subject is able to jog in a straight line
Lower Extremity Functional Scale (LEFS) | measured at PT Evaluation and 24th visit or 12 weeks Post-op (if missed appointments)
  All subjects will complete the LEFS questionnaire which contains 20 questions about a person's ability to perform everyday tasks. The maximum possible score is 80 points, indicating very high function. The minimum possible score is 0 points, indicating very low function.
Brief Resiliency Scale | measured at PT Evaluation and 24th visit or 12 weeks Post-op (if missed appointments)
  All subjects will complete the Brief Resiliency Scale which assesses the ability to bounce back. The possible score range is from 1 (low resilience) to 5 (high resilience)
Norwich Patellar Instability | measured at PT Evaluation and 24th visit or 12 weeks Post-op (if mised appointments)
  MPFL reconstruction subjects will complete the Norwich Patellar Instability which assesses patellar instability symptoms. The score is made up of 0 to 250. The total score is then converted to a percentage based on the number of scored responses. A higher percentage up to maximum 100% indicates the severity of patellar instability.
2000 IKDC Subjective Knee Evaluation Form | measured at PT Evaluation and 24th visit or 12 weeks Post-op (if missed appointments)
  ACL reconstruction patients with complete the 2000 IKDC Subjective Knee Evaluation Form. The IKDC is a patient-completed tool, which contains sections on knee symptoms (7 items), function (2 items), and sports activities (2 items). Scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms)

SECONDARY OUTCOMES:
Discomfort level | Measured at each treatment follwoing each BFR exercise - Specific Aim 2
  Measurement subject report discomfort level following each BFR exercise
Effort Level | Measured at each treatment follwoing each BFR exercise - Specific Aim 2
  Measurement subject report effort level following each BFR exercise

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kentucky Sports Rehabilitation, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Undecided